CLINICAL TRIAL: NCT05372445
Title: MicrobiAr: Characterization and Follow-up of Microbiome and Health Indicators in Obese, Pre-Diabetes and Type 2 Diabetes Cohorts Undergoing a Plant-based Diet and Lifestyle Intervention
Brief Title: Microbiome and Health Indicators in People With Obesity, Prediabetes and Type 2 Diabetes Undergoing a Lifestyle Intervention
Acronym: MicrobiAr
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Council of Scientific and Technical Research, Argentina (Other Government)
Collaborators: Facultad de Ingeniería - Universidad Austral (Unknown); Instituto de Inmunología, Genética y Metabolismo (INIGEM, CONICET-UBA) (Unknown); Illumina, Inc. (Industry); Zymo Research (Unknown); Instituto de Investigación y Desarrollo en Bioingeniería y Bioinformática (IBB, CONICET-UNER) (Unknown)
Responsible Party: Principal Investigator, Juan Pablo Bustamante, Bioinformatician, PhD in Biological Chemistry, National Council of Scientific and Technical Research, Argentina
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MicrobiAr
Record Dates: First submitted 2022-05-08; First posted 2022-05-12 (Actual); Last update posted 2022-08-01 (Actual); Status verified 2022-07

CONDITIONS: Diabetes Mellitus, Type 2; Obesity; PreDiabetes
Keywords: microbiota; microbiome; plant-based diet; type 2 diabetes remission; metabolic syndrome; caloric restriction; metabolic pathways
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Obesity; Prediabetic State; Metabolic Syndrome

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- Reference Group (No Intervention): People between 30-60 years old, without obesity, prediabetes or type 2 diabetes.
  The purpose of this group is to characterize gut microbiota and microbiome to set the reference values of the argentinian local population.
- Obesity Group A (Active Comparator): People between 30-60 years old, diagnosed with obesity assigned to the non-intensive intervention.
  Interventions: Behavioral: Non-intensive intervention
- Obesity Group B (Experimental): People between 30-60 years old, diagnosed with obesity assigned to the intensive intervention.
  Interventions: Behavioral: Intensive intervention
- Prediabetes Group A (Active Comparator): People between 30-60 years old, diagnosed with prediabetes assigned to the non-intensive intervention.
  Interventions: Behavioral: Non-intensive intervention
- Prediabetes Group B (Experimental): People between 30-60 years old, diagnosed with prediabetes assigned to the intensive intervention.
  Interventions: Behavioral: Intensive intervention
- Type 2 Diabetes Group A (Active Comparator): People between 30-60 years old, diagnosed with type 2 diabetes assigned to the non-intensive intervention.
  Interventions: Behavioral: Non-intensive intervention
- Type 2 Diabetes Group B (Experimental): People between 30-60 years old, diagnosed with type 2 diabetes assigned to the intensive intervention.
  Interventions: Behavioral: Intensive intervention

INTERVENTIONS:
Behavioral: Non-intensive intervention — After an evaluation of 7 day initial food-recall, subjects will receive counseling in order to improve their dietary habits, according to the American Diabetes Association 2019 Guidelines. The goals of this intervention are (i) achieve a caloric restriction of 500 kcal from their habitual energy intake, (ii) prioritize natural, minimally processed foods with a low glycemic index and glycemic load, (iii) eat lean protein sources, both from plant and animal origin and (iv) gradual increments of fiber intake, to achieve at least the minimum recommendations for the general population.
  The frequency of the follow-up appointments will be every 4 weeks, alternating between a clinical control and nutritional one. Therefore, the planned nutritional follow-up frequency will be every 2 months. In these appointments, the objective will be to achieve the mentioned energy intake reduction of 500 kcal, aiming to the nutritional goals previously mentioned, with the aid of the food-recalls.
  Other Names: Group A
  Arms: Obesity Group A; Prediabetes Group A; Type 2 Diabetes Group A
Behavioral: Intensive intervention — People will have virtual education with food and nutrition coaching workshops, as well as weekly meetings in small groups as a support and follow-up groups. The frequency of the face-to-face follow-up appointments will be every 3 weeks.
  The nutritional intervention will emphasize the consumption of mainly minimally processed food from plant origin. A vitamin b12 supplement per week will be provided. This intervention group will have 2 stages. First stage will have a duration of 3 months setting the nutritional bases going to a plant-based diet with basic considerations regarding fiber intake reducing meat consumption, and incorporating protein from vegetable sources, among other considerations. Second stage will progress to higher levels of fiber and others nutritional requeriments in order to intensify the nutritional plant-based intervention.
  Other Names: Group B
  Arms: Obesity Group B; Prediabetes Group B; Type 2 Diabetes Group B

SUMMARY:
The incidence of type 2 diabetes worldwide is growing rapidly, being one of the fastest growing global health emergencies of the 21st century according to the International Diabetes Federation. In MicrobiAr the investigators seek to achieve type 2 diabetes remission through a plant-based diet and lifestyle intervention identifying and characterizing key changes on the gut microbiome during clinical transitions. Specifically, the investigators aim to characterize and follow-up metabolic pathways from gut microbiome and how they evolve as long as health indicators do over the 2 years of this study.

DETAILED DESCRIPTION:
The present study has 2 stages, one cross-sectional and the other longitudinal. In the cross-sectional stage, a characterization of a single sampling of 480 people divided into 4 cohorts of 120 people each will be carried out: reference controls, subjects with obesity, with prediabetes and with type 2 diabetes. A clinical history will be made, as long as a 7-day food record and clinical laboratory tests. Anthropometric assessment will be carried out by recording weight, height, waist and hip circumference, determination of waist/hip ratios, as well as taking 4 skinfolds, bicipital, triceps, subscapular and suprailiac, arm and calf measurements and force through a dynamometer. The 480 people will also undergo gut microbiota and microbiome tests from stool samples.

During the longitudinal stage, subjects of each cohort (120 with obesity, 120 with prediabetes and 120 with type 2 diabetes) will be randomly divided into two intervention groups (with 60 subjects each). One group will follow a non-intensive intervention (personalized face-to-face follow-up every 2 months). The other group will follow an intensive intervention (personalized face-to-face follow-up every 3 weeks and a weekly remote group meeting). In both cases, a food plan will be followed based on the recommendations of the nutrition service of the Hospital de Clínicas, Argentina, in accordance with recommendations from the American Diabetes Association (ADA) 2019 guidelines with an emphasis on plant-based diet and whole foods.

Follow-up and nutritional guidance

Groups of 15 subjects from each intervention arm will be led by 3 healthcare professionals. In every case, the group's functions will be:

1. Obtain a unique 7 day food-recall from all subjects, and upload the data to "MAR24" platform (for the transversal stage).
2. Obtain a 2 day food-recall (including one day from the weekend) from all subjects every two months, and upload the data to "MAR24" platform (for the longitudinal stage).
3. Complete a shared spreadsheet with clinical, biochemical and anthropometric parameters of every subject's visits to the hospital.
4. Collaborate in Whatsapp unidirectional groups. In the non-intensive arm, the messages will only be to remember patients about their visits to the hospital, while in the intensive arm it will also be about other activities, such as workshops.
5. Detect subjects who miss their appointments, to establish personalized contact and apply motivational strategies in order to reduce dropout risk.

To accomplish the mentioned tasks, the group leaders will have support from several students from nutrition careers and healthcare professionals.

Influence of physical activity and exercise

A structured physical exercise protocol will be delivered to all subjects. This protocol includes a warm-up, 3 series of 1 minute of eight different strength exercises, with 2 a minute rest. The objective is to accomplish three sessions per week, which can be done in person and supervised by specialists in the Hospital, or online via video call. Subjects will have to record the amount of achieved repetitions in each series of every exercise already done by each session.

The training volume will be adapted according to the subject's capabilities and progress, with the objective of increasing the number of series and reducing resting time between exercises.

Specific follow-up and support proposals for the intensive intervention

In addition to the already mentioned tasks in the follow-up and nutritional guidance's section, for the intensive intervention subjects, group's functions will also be:

1. Collaborate in the assembly and execution of virtual food education workshops;
2. Coordinate weekly meetings with the 15 assigned subjects, where adherence should be encouraged during the first 3 months. Then, meetings will be spaced out at a minimum of 15 days to 30 days;
3. Contribute to the planning of various activities that seek to maximize adherence to the clinical trial of the entire intensive intervention group;
4. Coordinate face-to-face visits for nutritional support every 3 weeks for each subject;
5. Monitoring adherence through 48-hour records (1 day a week and 1 day a weekend) using the MAR24 platform. Data will be collected by phone calls or video calls to each subject with a frequency of 1 call per month.

ELIGIBILITY:
Inclusion Criteria for control or reference group:

* Subjects without type 2 diabetes, obesity, prediabetes (glucose intolerance), or metabolic syndrome
* HbA1c less than 42mmol/mol (<5.7%)
* BMI between 18.5 and 24.9

Inclusion Criteria for people with obesity:

* BMI greater than 30

Inclusion Criteria for people with prediabetes:

* Fasting glucose between 110 and 125 mg/dl
* HbA1c between 42 and 47 mmol/mol (5.7% to 6.4%)
* BMI greater than 30

Inclusion Criteria for people with type 2 diabetes:

* Fasting glucose > 126 mg/dl
* HbA1c > 48mmol/mol (6.5% or higher)
* BMI greater than 30
* Treatment with metformin at therapeutic dose (1500-2000 mg/day) or maximum tolerated dose.

Exclusion Criteria:

* Subjects with obesity, pre-diabetes medicated with metformin or another drug for diabetes or obesity
* Subjects with type 2 diabetes medicated with another drug that is not metformin
* Subjects with type 2 diabetes diagnosed over 6 years
* Subjects with type 2 diabetes requiring insulin
* Chronic kidney disease grade greater than 3 (measured by EPI)
* Subjects with type 1 diabetes
* Intestinal diseases, Crohn's, ulcerative colitis, celiac disease
* Use of antibiotics in the last 3 months
* Pregnancy, lactation
* Psychiatric disorders
* Eating disorder
* Gastric bypass surgery
* Transplanted people
* Oncological pathology diagnosed less than 5 years
* Subjects who do not wish to sign the informed consent
* Subjects who do not agree to participate in the study over the 2 years follow-up
* Subjects who do not have electronic devices and the internet to hold virtual meetings

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 480 (Estimated)
Dates: Start 2022-05-30 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Clinical improvements in people with type 2 diabetes, prediabetes, or obesity | at 2 years, checked every 6 months
  These clinical improvements will be defined as:
  1. In the group of subjects with type 2 diabetes, remission to non-diabetic stage. Considering remission as measuring HbA1c values lower than 6,5% at least 6 months after beginning the lifestyle intervention and 3 months after cessation of any pharmacotherapy, according to the "Consensus Report: Definition and Interpretation of Remission in Type 2 Diabetes", Diabetes Care 2021;44(10):2438-2444.
  2. In the group of subjects with prediabetes, remission to normal glycemia / HbA1c values. Considering normal glycemia lower than 100 mg/gl and HbA1c lower than 5.7%.
  3. In the group of overweight-obese subjects, a 10% decrease in weight compared to baseline weight, maintained during the second year of follow-up.
  Any of the three possible situations will be considered as a clinical improvement event.
Gut microbiota metabolic pathways changes | at 2 years, checked every 6 months
  Increase in the number of gut microbiota metabolic pathways possibly expressed in subjects of intensive intervention compared to their baseline states and also compared to subjects of the non-intensive intervention. This metric refers to possibly expressed metabolic pathways predicted from shotgun metagenomics analysis related to regulation of inflammatory processes, carcinogenesis, intestinal barrier function, oxidative stress, production of SCFAs, regulation of immune response and inflammation, production of derivative aromatic amino acids, regulation of bile acids (synthesis of derivative metabolites of cholesterol), regulation of the level of phospholipid synthesis (anaerobic metabolism of choline).

SECONDARY OUTCOMES:
Metabolic syndrome regression | at 2 years, checked every 6 months
  Participants with diagnosis of metabolic syndrome at baseline who no longer meet metabolic syndrome criteria, according to those established by the Joint Interim Statement in 2009 (Harmonizing the metabolic syndrome: a joint interim statement of the International Diabetes Federation Task Force on Epidemiology and Prevention; National Heart, Lung, and Blood Institute; American Heart Association; World Heart Federation; International Atherosclerosis Society; and International Association for the Study of Obesity. Circulation. 2009;120:1640 -1645.)
Insulin resistance | at 2 years
  Measured by HOMA-IR, HOMA-B or triglyceride: HDL-C ratio.
Gut microbiota diversity changes | at 2 years, checked every 6 months
  Increase of diversity in gut microbiota observed in subjects of the intensive intervention compared to subjects of the non-intensive intervention and also compared to their baseline states.

CONTACTS AND LOCATIONS:
Overall Officials: Juan Bustamante, PhD, Principal Investigator — CONICET Researcher; Gustavo Frechtel, PhD, Principal Investigator — CONICET Researcher
Locations (1):
- Hospital de Clínicas "José de San Martín", Capital Federal, Buenos Aires, Argentina

IPD SHARING:
Plan to Share IPD: Yes
all required data in order to reproduce the publication
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: starting immediately after publication in a peer reviewed journal
Access Criteria: all required data in order to reproduce the publication will be full available in our website www.microbiar.com through a specific section that will be implemented for this aim.

REFERENCES:
- [Background] Alberti KG, Eckel RH, Grundy SM, Zimmet PZ, Cleeman JI, Donato KA, Fruchart JC, James WP, Loria CM, Smith SC Jr; International Diabetes Federation Task Force on Epidemiology and Prevention; Hational Heart, Lung, and Blood Institute; American Heart Association; World Heart Federation; International Atherosclerosis Society; International Association for the Study of Obesity. Harmonizing the metabolic syndrome: a joint interim statement of the International Diabetes Federation Task Force on Epidemiology and Prevention; National Heart, Lung, and Blood Institute; American Heart Association; World Heart Federation; International Atherosclerosis Society; and International Association for the Study of Obesity. Circulation. 2009 Oct 20;120(16):1640-5. doi: 10.1161/CIRCULATIONAHA.109.192644. Epub 2009 Oct 5. PMID 19805654
- [Background] Riddle MC, Cefalu WT, Evans PH, Gerstein HC, Nauck MA, Oh WK, Rothberg AE, le Roux CW, Rubino F, Schauer P, Taylor R, Twenefour D. Consensus Report: Definition and Interpretation of Remission in Type 2 Diabetes. Diabetes Care. 2021 Aug 30;44(10):2438-44. doi: 10.2337/dci21-0034. Online ahead of print. PMID 34462270